CLINICAL TRIAL: NCT04059705
Title: The Impact of Dual-task Training on Attention and Motor Function in Older Adults With Mild Cognitive Impairment
Brief Title: Dual-task Training for Function in MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Nikhil Satchidanand, Assistant Professor of Medicine, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003525
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment
Keywords: motor function; cognitive; attention; dual-task; physical activity; cognition; older adult; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study utilizes a one-group design with repeated measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-Task Intervention (Experimental): This study arm will receive the dual-task training program.
  Interventions: Behavioral: Dual-Task Training

INTERVENTIONS:
Behavioral: Dual-Task Training — The ThinkFIT intervention will involve two days per week participation in simultaneous cognitive and motor training activities, facilitated by the SMARTFit Multisensory FItness System.
  Other Names: ThinkFIT Intervention, SMARTFit Multisensory Fitness System

SUMMARY:
Mild cognitive impairment (MCI) is an intermediate stage between the expected cognitive decline of normal aging and severe dementia associated with Alzheimer's disease (AD). In the United States about 20% of older adults have MCI. Loss of cognitive function in aging can have far-reaching and devastating impacts on functional status, independence, and quality of life. Unfortunately, the therapeutic options to slow progression of cognitive decline in aging are limited. Dual-task training; that which involves simultaneous cognitive and motor challenges, is a high-impact potential therapy to slow progressive loss of both motor and cognitive function in aging. The purpose of this trial is to examine the feasibility and therapeutic impact of a novel dual-task physical activity intervention on executive and motor functions among adults, 65 years or older, who have MCI. the investigative team anticipates that findings from this trial will inform development of larger community-based studies focused on improving function and ability to maintain independence in older age.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is an intermediate stage between the expected cognitive decline of normal aging and severe dementia associated with Alzheimer's disease (AD). In the United States about 20% of older adults have MCI, and approximately 15% per year of those with MCI will progress to AD. With our rapidly aging society, we are approaching a public health crisis for which we are not fully prepared. Impaired cognitive function in aging can have far-reaching and devastating impacts on functional status, ability to maintain independence, and overall quality of life. Unfortunately, the therapeutic options to slow progression of cognitive decline in aging are limited.

Dual-task training that involves simultaneous cognitive and motor challenges improves certain domains of both cognitive and motor function in older adults with MCI. However, we do not yet know the optimal methods of delivering this high-impact potential therapy in community-based settings with unique limitations and strengths. Therefore, the aims are to; 1) test the feasibility of conducting a community-based dual-task (thinking while exercising) physical activity intervention among adults, 65 years or older, with MCI; and 2) examine the impact of dual-task training on attention and motor function among adults, 65 years or older, with MCI.

To accomplish these aims the investigators will conduct an 12-week, dual-task training program using the SmartFit Multisensory Fitness System (Oxnard, CA) among older adults with MCI. Our group-based training program involves two 1-hour training sessions per week, designed to simultaneously engage the mind and body, while promoting self-efficacy. Attention and motor function will be assessed prospectively.

The investigators anticipate that findings from this trial will inform development of methods to bring evidence-based, non-invasive therapies into communities in need, in order to preserve function, independence, and quality of life well into older age.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Male or female
* Mild (23 - 26 points) cognitive impairment as screened by the Montreal Cognitive Assessment
* Having no absolute contraindications to non-physician supervised exercise as guided by the American College of Sports Medicine and Centers for Disease Control and Prevention.

Exclusion Criteria:

* Having any condition that prevents safe participation in non-physician supervised exercise as screened using the Physical Activity Readiness Questionnaire for Older Adults
* Blood pressure >180 mmHg systolic or 100 mmHg diastolic at baseline
* Presence of severe illness or disability
* Lower body amputation
* Cognitive Impairment beyond mild level, preventing provision of informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Motor Function from baseline to 12 weeks | baseline, week 6, week 12
  Change in motor function will be assessed prospectively using the Short Physical Performance Battery.
Change in Attention from baseline to 12 weeks | baseline, week 6, week 12
  Attention will be assessed prospectively using the Stroop Task and Trail-making Test.

SECONDARY OUTCOMES:
Change in Exercise Self Efficacy from baseline to 12 weeks | baseline, week 12
  Self efficacy for exercise will be assessed using the Self Efficacy for Exercise Scale. Total score is derived by summing the individual scores for each question. Scoring range for this instrument is 0 - 90 points with higher scores representing better outcomes.
Outcome Expectations for Exercise from baseline to 12 weeks | baseline, week 12
  Outcome Expectations for exercise will be assessed using the Outcome Expectations for Exercise Scale. This instrument has 9 total items. Total score is derived by summing the responses to these items and dividing by the number of responses. Scoring is out of 9 points, with higher scores demonstrating higher outcomes expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Satchidanand, PhD, Principal Investigator — University at Buffalo, State University of New York
Locations (1):
- Buffalo-Niagara YMCA, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will allow data and supportive documents to be available to users only under a defined data-sharing agreement that enforces (a) their commitment to using the data only for research purposes and does not identify any individual research participant; (b) the commitment to secure all research data using appropriate technology; (c) prohibition of redistribution of the data to third parties, as well as proper acknowledgement of the data resource, and (d) a commitment to destroying and/or returning the data after analyses have been completed. De-identified data will be maintained on a University at Buffalo server and will be shared via encrypted devices. Co-Investigators may access the data collected as part of their aims. Investigators working on the project will have access to the data only through the principal investigator. The data will be monitored routinely to maintain security, safety, and productivity.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1-year after first publication
Access Criteria: Final data sets will be made available upon specific request and under an authorized Data Use Agreement. This, in addition to the publications being made available via PubMed Central, will enable validation of results by recipients.